CLINICAL TRIAL: NCT00963937
Title: A Randomized, Multicenter, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Oral Sumatriptan for the Acute Treatment of Migraine in Children and Adolescents
Brief Title: Study to Evaluate the Efficacy and Safety of Oral Sumatriptan for the Acute Treatment of Migraine in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111035
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-06

CONDITIONS: Migraine Disorders
Keywords: adolescent; sumatriptan; children; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sumatriptan 25 mg (Active Comparator)
  Interventions: Drug: Sumatriptan 25 mg
- Sumatriptan 50 mg (Active Comparator)
  Interventions: Drug: Sumatriptan 50 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sumatriptan 25 mg — One Sumatriptan 25mg tablet and one Matching Placebo tablet should be administered as soon as possible (within 30 minutes) after the development of a migraine associated with 3 or more pain on a 5-grade scale.
  Arms: Sumatriptan 25 mg
Drug: Sumatriptan 50 mg — Two Sumatriptan 25mg tablets should be administered as soon as possible (within 30 minutes) after the development of a migraine associated with 3 or more pain on a 5-grade scale.
  Arms: Sumatriptan 50 mg
Drug: Placebo — Two Matching Placebo tablets should be administered as soon as possible (within 30 minutes) after the development of a migraine associated with 3 or more pain on a 5-grade scale.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a range of doses of oral sumatriptan for the acute treatment of migraine in children ages 10 to 17.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >10 years of age and <17 years of age at the informed consent and the Randomization Visit.
* Subject has migraine with or without aura (ICHD-II criteria, 1.1 or 1.2.1). A minimum of a six month history of migraine prior to entry into the study is required.
* Subject has a history of at least two, but no more than eight, attacks per month for the two months prior to entry into the study.
* All migraine attacks associated with 3 or more pain on a 5-grade scale should last a minimum of three hours for the two months prior to entry into the study.
* Subject has shown nonresponse to at least one NSAIDs or acetaminophen for the two months prior to entry into the study.
* Subject is able to distinguish migraine from other headaches (e.g., tension-type headache).
* Subject is able to read, comprehend, and complete subject diaries.
* Males or female subjects. Female subjects are eligible for participation in the study if they are one of the following
* Females of non-childbearing potential (i.e., physiologically incapable of becoming pregnant or have undergone female sterilization)
* Females of childbearing potential, and who have a negative pregnancy test at the Screening Visit, and agree to use one of the following GlaxoSmithKline (GSK)-specified highly effective methods for avoiding pregnancy:
* Abstinence
* Oral Contraceptive, either combined or progestogen alone
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject)
* Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository)
* Subject's parent or legal guardian is willing and able to provide informed consent prior to subject entry into the study.
* Subject is willing and able to provide informed assent prior to entry into the study.
* Subjects considered for enrolment must have a QTc (either QTc B (Bazett's correction) or QTc F (Fridericia's correction)) <450msec at the Screening Visit, with the exception of subjects with bundle branch block (for whom either QTc B or QTc F must be <480msec).

Note: For the purposes of these criteria, QTc B is defined as (QT interval msec) / (square root of RR interval seconds); and QTc F is defined as (QT interval msec) / (cube root of RR interval seconds).)

* Liver function test at the Screening Visit: AST and ALT <2xULN; alkaline phosphatase and total bilirubin <1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)

Exclusion Criteria:

* Subject is < 30 kg.
* Subject has 15 or more headache days per month in total (migraine, probable migraine, or tension-type). Subject has retinal (ICHD-II 1.4), basilar (ICHD-II 1.2.6), hemiplegic (ICHD-II 1.2.4 or 1.2.5), or Ophthalmoplegic migraine (ICHD-II 13.17). Subject has secondary headaches.
* Subject has a history of cerebrovascular disease or ischemic cerebrovascular disease.
* Subject has a history of myocardial infarction.
* Subject has uncontrolled hypertension.
* Subject has symptoms or signs of ischemic cardiac syndromes.
* Subject has variant angina.
* Subject has evidence of a peripheral vascular syndrome.
* Subject has evidence or history of epilepsy or structural brain lesions which lower the convulsive threshold, or has been treated with an antiepileptic drug for seizure control.
* Subject has a history of impaired hepatic or renal function that, in the investigator (or subinvestigator)'s opinion, contraindicates participation in this study. Subject has unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice). Subject has cirrhosis. Subject has known biliary abnormalities (with the exception of Gilberts's syndrome or asymptomatic gallstones).
* Subject has hypersensitivity, allergy, intolerance, or contraindication to the use of any triptan (including all sumatriptan preparations) or sulfonamide compounds.
* Subject has used an ergot medication in the previous three months for migraine prophylaxis or is taking a medication that is not stabilized (i.e., change of dose within the past 2 months) for either chronic or intermittent migraine prophylaxis.
* Subject has taken, or plans to take, a monoamine oxidase inhibitor (MAOI) anytime within the two weeks prior to entry into the study.
* Subject has evidence of psychotropic, alcohol, or substance abuse within the last year.
* Subject has participated in any investigational drug trial within the previous 3 months or plans to participate in another study at any time during this study.
* Subject has any concurrent medical or psychiatric condition which, in the investigator (or subinvestigator)'s judgment, contraindicates participation in this clinical trial.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2009-09-28; Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants took 2 tablets of placebo matched to sumatriptan 25 milligrams (mg) within 30 minutes after the development of a migraine associated with a score of 3 or more for pain on a 5-grade, self-rating scale to assess the pain intensity of a migraine: 1 = none, 2 = mild, 3 = mild to moderate, 4 = moderate to severe, and 5 = severe.
- Sumatriptan 25 mg: Participants took 1 tablet of sumatriptan 25 mg and 1 tablet of placebo matched to sumatriptan 25 mg within 30 minutes after the development of a migraine associated with a score of 3 or more for pain on the 5-grade scale.
- Sumatriptan 50 mg: Participants took 2 tablets of sumatriptan 25 mg within 30 minutes after the development of a migraine associated with a score of 3 or more for pain on the 5-grade scale.
Period: Overall Study
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg
Started | 89 | 44 | 45
Completed | 70 | 33 | 41
Not Completed | 19 | 11 | 4
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Physician Decision | 18 | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Total
Number analyzed (Participants) | 70 | 33 | 41 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in the Full Analysis Set (FAS), comprised of all participants who took at least one dose of investigational product (IP) and provided any post-treatment efficacy assessment. Participants who withdrew from the study before completion did not receive IP and thus contributed no baseline data.
  Years | 13.9 (2.04) | 14.5 (2.18) | 14.1 (1.96) | 14.1 (2.05)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected in the Full Analysis Set (FAS), comprised of all participants who took at least one dose of investigational product (IP) and provided any post-treatment efficacy assessment. Participants who withdrew from the study before completion did not receive IP and thus contributed no baseline data.
  Participants
    Female | 39 | 17 | 28 | 84
    Male | 31 | 16 | 13 | 60
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in the Full Analysis Set (FAS), comprised of all participants who took at least one dose of investigational product (IP) and provided any post-treatment efficacy assessment. Participants who withdrew from the study before completion did not receive IP and thus contributed no baseline data.
  participants | 70 | 33 | 41 | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reported Pain Relief at 120 Minutes Post-Treatment
Description: Pain relief was defined as at least a 2-grade reduction in pain intensity on a 5-grade scale in participants who had not used headache rescue medication before assessment. A pain intensity score of 5 was assigned for all subsequent assessments if a participant took rescue medication (a single oral dose for the treatment of migraine pain or associated symptoms). The 5-grade scale is a participant's self-rating scale to assess the pain intensity of a migraine with the following scores: 1 = none, 2 = mild, 3 = mild to moderate, 4 = moderate to severe, and 5 = severe.
Time Frame: 120 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: Full Analysis Set (FAS): all participants in the Safety Population (all participants who took >=1 dose of investigational product [IP]) who provided any post-treatment efficacy assessment. Analysis was performed on the last observation carried forward (LOCF) dataset (imputed by LOCF method). Only post-treatment values were used for imputation.
Measure: Number; unit: percentage of participants
Groups:
- Sumatriptan Pooled: All participants receiving either sumatriptan 25 mg or 50 mg
Arm/Group | Placebo | Sumatriptan Pooled
Number analyzed (Participants) | 70 | 74
percentage of participants | 38.6 | 31.1
Statistical Analysis 1: Comparison: Placebo vs Sumatriptan Pooled; Test type: Superiority or Other; p = 0.345, Chi-squared — Multiplicity was not considered because the primary analysis included a single statistical comparison; Percent Difference = -7.49, 95% CI 2-sided [-23.02 to 8.04] — Percent difference = sumatriptan pooled group minus the placebo group

2. Secondary Outcome: Percentage of Participants Who Reported Pain Relief at 30, 60, 120, and 240 Minutes Post-Treatment
Description: as for outcome 1
Time Frame: 30, 60, 120, and 240 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: FAS. The analysis was performed on the LOCF dataset.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Number analyzed (Participants) | 70 | 33 | 41 | 74
percentage of participants
  30 minutes post-treatment | 4.3 | 0 | 9.8 | 5.4
  60 minutes post-treatment | 18.6 | 9.1 | 7.3 | 8.1
  120 minutes post-treatment | 38.6 | 33.3 | 29.3 | 31.1
  240 minutes post-treatment | 51.4 | 66.7 | 61.0 | 63.5

3. Secondary Outcome: Percentage of Participants Who Were Pain Free at 30, 60, 120, and 240 Minutes Post-Treatment
Description: Pain free was defined as a post-treatment pain intensity score of 1 on a 5-grade scale in participants who had not used headache rescue medication before assessment. A pain intensity score of 5 was assigned for all subsequent assessments if a participant took a rescue medication. The 5-grade scale is a participant's self-rating scale to assess the pain intensity of a migraine with the following scores: 1 = none, 2 =mild, 3=mild to moderate, 4=moderate to severe, and 5=severe.
Time Frame: 30, 60, 120, and 240 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: FAS. The analysis was performed on the LOCF dataset.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Number analyzed (Participants) | 70 | 33 | 41 | 74
percentage of participants
  30 minutes post-treatment | 2.9 | 0 | 2.4 | 1.4
  60 minutes post-treatment | 12.9 | 3.0 | 2.4 | 2.7
  120 minutes post-treatment | 28.6 | 24.2 | 19.5 | 21.6
  240 minutes post-treatment | 47.1 | 63.6 | 39.0 | 50.0

4. Secondary Outcome: Percentage of Participants Who Were Photophobia Free at 30, 60, 120, and 240 Minutes Post-Treatment
Description: Photophobia (sensitivity to light) is one of the associated symptoms of a migraine. A participant was assessed as photophobia free when the symptom was recorded as "absent" at each time point in his or her patient diary. Photophobia was recorded as "present" for all subsequent assessments if a participant took rescue medication.
Time Frame: 30, 60, 120, and 240 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: FAS. The analysis was performed on the LOCF dataset. Only participants who had photophobia at the time of treatment were included in the denominator.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Number analyzed (Participants) | 36 | 15 | 13 | 28
percentage of participants
  30 minutes post-treatment | 16.7 | 13.3 | 15.4 | 14.3
  60 minutes post-treatment | 44.4 | 26.7 | 38.5 | 32.1
  120 minutes post-treatment | 52.8 | 60.0 | 46.2 | 53.6
  240 minutes post-treatment | 69.4 | 80.0 | 69.2 | 75.0

5. Secondary Outcome: Percentage of Participants Who Were Phonophobia Free at 30, 60, 120, and 240 Minutes Post-Treatment
Description: Phonophobia (sensitivity to sound) is one of the associated symptoms of a migraine. A participant was assessed as phonophobia free when the symptom was recorded as "absent" at each time point in his or her patient diary. Phonophobia was recorded as "present" for all subsequent assessments if a participant took rescue medication.
Time Frame: 30, 60, 120, and 240 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: FAS. The analysis was performed on the LOCF dataset. Only participants who had phonophobia at the time of treatment were included in the denominator.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Number analyzed (Participants) | 22 | 14 | 16 | 30
percentage of participants
  30 minutes post-treatment | 22.7 | 50.0 | 12.5 | 30.0
  60 minutes post-treatment | 45.5 | 57.1 | 25.0 | 40.0
  120 minutes post-treatment | 63.6 | 64.3 | 43.8 | 53.3
  240 minutes post-treatment | 72.7 | 78.6 | 68.8 | 73.3

6. Secondary Outcome: Percentage of Participants Who Were Nausea Free at 30, 60, 120, and 240 Minutes Post-Treatment
Description: Nausea is one of the associated symptoms of a migraine. A participant was assessed as nausea free when the symptom was recorded as "absent" at each time point in his or her patient diary. Nausea was recorded as "present" for all subsequent assessments if a participant took rescue medication.
Time Frame: 30, 60, 120, and 240 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: FAS. The analysis was performed on the LOCF dataset. Only participants who had nausea at the time of treatment were included in the denominator.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Number analyzed (Participants) | 21 | 10 | 8 | 18
percentage of participants
  30 minutes post-treatment | 47.6 | 40.0 | 12.5 | 27.8
  60 minutes post-treatment | 66.7 | 40.0 | 12.5 | 27.8
  120 minutes post-treatment | 81.0 | 70.0 | 50.0 | 61.1
  240 minutes post-treatment | 81.0 | 70.0 | 50.0 | 61.1

7. Secondary Outcome: Percentage of Participants Who Were Free of Vomiting at 30, 60, 120, and 240 Minutes Post-Treatment
Description: Vomiting is one of the associated symptoms of a migraine. A participant was assessed as being free of vomiting when the symptom was recorded as "absent" at each time point in his or her patient diary. Vomiting was recorded as "present" for all subsequent assessments if a participant took a rescue medication.
Time Frame: 30, 60, 120, and 240 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: FAS. The analysis was performed on the LOCF dataset. Only participants who had vomiting at the time of treatment were included in the denominator.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Number analyzed (Participants) | 0 | 1 | 0 | 1
percentage of participants
  30 minutes post-treatment |  | 0 |  | 0
  60 minutes post-treatment |  | 0 |  | 0
  120 minutes post-treatment |  | 100.0 |  | 100.0
  240 minutes post-treatment |  | 100.0 |  | 100.0

8. Secondary Outcome: Percentage of Participants Who Used Rescue Medication Between the Time of Dosing and 240 Minutes Post-Treatment
Description: Rescue medication included one of the following: a single oral dose of a nonsteroidal anti-inflammatory drug (NSAID) or acetaminophen, not to exceed the maximum recommended single dose; and anti-emetics (a drug to prevent vomiting).
Time Frame: within 240 minutes post-treatment (Randomization through Final Visit [Week 6])
Population: FAS. The analysis was performed on the observed case dataset, a dataset without any imputation of missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Number analyzed (Participants) | 70 | 33 | 41 | 74
percentage of participants | 12.9 | 12.1 | 14.6 | 13.5

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs) and non-serious AEs were collected from the start of IP through follow-up contact (6 weeks plus or minus 7 days).
Arm/Group | Placebo | Sumatriptan 25 mg | Sumatriptan 50 mg | Sumatriptan Pooled
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/33 | 0/41 | 0/74
Other Adverse Events (participants affected / at risk) | 5/70 | 2/33 | 3/41 | 5/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=70) | Sumatriptan 25 mg (N=33) | Sumatriptan 50 mg (N=41) | Sumatriptan Pooled (N=74)
Blood creatine phosphokinase increased (Investigations) | 4 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 3 | 3
Somnolence (Nervous system disorders) | 1 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.